CLINICAL TRIAL: NCT07269964
Title: At-home tDCS as Maintenance Therapy Following Successful Treatment With rTMS, ECT, and Esketamine - A Pilot Study
Brief Title: At-Home tDCS as Maintenance Therapy
Acronym: MaintenanceDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Ulrike Vogelmann, Dr.med., Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RWNM_tDCS_Maintenance
Record Dates: First submitted 2025-09-08; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: MDD; Severe Depression; Major Depressive Episode
Keywords: Non Invasive Brain Stimulation (NIBS); tDCS; at-home treatment; tdcs at home; transcranial direct current stimulation
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Single arm, pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- at home tdcs after ECT, rTMS or Esketamine treatment (Active Comparator): Transcranial Direct Current Stimulation (tDCS) at home, 20 sessions, 2mA (5 days/week, for 4 weeks) as at home maintenance treatmentafter successfull ECT, rTMS or Esketamine treatment.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Description: Transcranial Direct Current Stimulation delivered at an intensity of 2 mA over electrodes at F3/F4 (bifrontal, over DLPFC), for 30 minutes a day, Monday to Friday, for a total 20 sessions.

SUMMARY:
The primary purpuse of this pilot study is to find out whether a home-based transcranial direct current stimulation (tDCS) program is feasible and well tolerated as maintenance therapy and whether there are early signs that it helps maintain the clinical clinical benefits achieved during successful acute inpatient treatment.

Participant population:

Adults (18+) with depressive disorder who had already improved/stabilized after acute treatment at our clinic (esketamine, repetitive transcranial magnetic stimulation , or electroconvulsive therapy).

Main questions:

Feasibility: Do participants reliably complete the home program and stay in the study?

Preliminary effectiveness: Do improvements of depressive symptoms hold up over the 4-week treatment and 2-week follow-up (based on self-report and clinician-rated scales)?

Participants receive standardized instruction from trained staff and a portable tDCS device (with cap and small sponge electrodes) and complete 20 home sessions over 4 weeks (5 per week), each 30 minutes at a very low current (2 mA); the device gently ramps current up/down for comfort.

During treatment, participants use a smartphone app with step-by-step guidance and reminders; sessions are automatically logged. They will also fill out short weekly self-rating questionnaires and join brief phone check-ins every 2 weeks.

Where:

Department and Outpatient Clinic of Psychiatry and Psychotherapy, Klinikum rechts der Isar, Technical University of Munich

Safety & data privacy:

The device monitors electrode contact and pauses automatically if contact is poor. Typical sensations can include mild tingling or redness. The app stores anonymized session data so the care team can track progress; no personal data are exchanged between the app and the stimulator, and access is via a secure clinical portal.

DETAILED DESCRIPTION:
Study type Open-label pilot clinical study.

Primary purpose To determine whether a home-based transcranial direct current stimulation (tDCS) maintenance program is feasible and well tolerated, and whether there are early signs that it helps maintain the clinical benefits achieved during successful acute inpatient treatment for depression.

Location Department and Outpatient Clinic of Psychiatry and Psychotherapy, Klinikum rechts der Isar, Technical University of Munich

Participants Adults (≥18 years) with a depressive disorder who already improved or stabilized after acute treatment in our hospital (such as esketamine, repetitive transcranial magnetic stimulation, or electroconvulsive therapy). Participants must be able to give informed consent. People in an acute crisis, with high suicide risk, or with medical reasons that make tDCS unsafe (e.g., certain implants near the head, significant skin disease at the electrode sites) are not included.

What is tDCS? tDCS uses a very low, constant electrical current delivered through two small sponge electrodes on a soft cap to gently modulate brain activity in areas linked to mood regulation. The at-home device ramps the current up and down gradually for comfort, and automatically pauses if contact with the skin is not adequate.

What participants will do Training & setup: Participants receive standardized instruction from trained staff and a portable tDCS device with a cap and sponge electrodes. Correct placement and skin preparation are well demonstrated.

Home treatment (4 weeks): 20 sessions (5 per week) at home, each 30 minutes at 2 mA. The device gives step-by-step prompts; current ramps up/down to improve comfort.

Check-ins & questionnaires:

Participants complete brief weekly questionnaires and have check-ins every 2 weeks. After finishing the 4-week program, there is a 2-week follow-up with a final assessment.

Usual care:

Ongoing medications or psychotherapy may continue unchanged and is not standardized in this pilot-study.

What the study measures:

Feasibility (primary objective): Is the at-home maintenance treatment after acute inpatient treatment well tolerated by patients? Improvements in MADRS and self reporting questionnaires as BDI-II.

Adherence:

How many of the 20 planned sessions each participant actually completes.

Safety:

Number and type of adverse events (AEs) and any device-related issues.

Preliminary effectiveness:

Whether maintenance or improvements hold up during treatment and follow-up are assessed using standardized self-rated and clinician-rated questionnaires.

Adverse effects:

Typical sensations can include mild tingling, redness, or a light headache; serious events are uncommon. Participants can pause or stop at any time and contact the team for support.

Data handling and privacy The app stores anonymized session data (e.g., time and completion of sessions) so the team can monitor progress.No personal identifiers are transmitted between the app and the stimulator. Access to study data is restricted to the clinical team via a secure portal.

Why this pilot matters Before running a large, controlled trial, we need to confirm that a home-based tDCS program is practical to deliver, acceptable to participants, and shows early signs of maintaining post-acute clinical benefits. Results from this pilot will guide decisions about a future randomized, posssibly sham-controlled study with a longer follow-up focused on relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Diagnosis according to ICD-10: recurrent depressive disorder, severe depressive disorder, schizoaffective disorder (depressive episode) or bipolar affective disorder (depressive episode).
* Clear indication for maintenance therapy after successful acute treatment (esketamine, rTMS, or ECT) with remission/improvement of symptoms.
* Capacity to provide informed consent, confirmed in a physician-led consent discussion.

Exclusion Criteria:

* Currently in the acute treatment phase of an affective disorder and non-response to previous treatments.
* Currently clinically relevant Axis II disorders.
* Suicidal risk, including suicidal ideation.
* Contraindications for tDCS: e.g., skin disease at electrode sites, cochlear implants.
* Neurological, somatic, or psychiatric comorbidities that could compromise validity or safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility, number of completed sessions | 4 weeks from baseline
  Feasibility:
  This is an open-label, single-arm pilot designed to determine whether a home-based tDCS maintenance program can be delivered reliably, safely, and acceptably after successful acute inpatient treatment. It's important to assess feasibility in order to observe whether participants can complete the 4-week, self-administered regimen with remote support and whether the procedure is well tolerated in a real-world home setting. Establishing feasibility is essential to ensure that a larger trial would be both deliverable and acceptable.
  Feasibility is determined by the number of tDCS sessions completed by patients. It is considered achieved at 75% protocol adherence, i.e., when 15 tDCS sessions are delivered.

SECONDARY OUTCOMES:
Depressive Symptoms assessed with MADRS | MADRS: Measured in week one, week two, week four during treatment phase and in week six during the follow up phase.
  Major Depression psychiatric symptoms assessed with the Montgomery Asberg Depression Rating Scale (MADRS). MADRS values are interpreted as follows: 0-6 = No depression, 07-19 = mild, 20-34 = moderate, 35-60 = severe.
  Outcome is the Difference in MADRS Score from baseline to post-treatment visit at week four and at week six (follow up phase)
BDI II | Measured at day 1 (baseline), week two (after completing ten at home sessions), week four(after completing full treatment) and followup at week 6.
  Major Depression psychiatric symptoms assessed with the Beck Depression Inventory (BDI-II). Outcome values are interpreted as follows: 0-13 = Minimal depression, 14-19 = Mild depression, 20-28 = Moderate depression, 29-63 = Severe depression
Safety based on the number of adverse events | Adverse events are monitored weekly: Baseline (pre-treatment), week 1, 2, 3, 4 and during follow up (week 6)
  Typical adverse events may include mild tingling or redness.
Analysis of monitored technical parameters | These parameters will be assessed daily during treatment period, i.e. tDCS treatment day 1-20 automatically
  Safety will be assessed not only by adverse events but also by device- and app-logged technical parameters that reflect safe delivery in the home setting. such as electrode-scalp contact quality as well as device/app error codes and battery-related interruptions; and the need for make-up sessions attributable to technical causes.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Technical University of Munich, TUM School of Medicine and Health, Department of Psychiatry and Psychotherapy, Munich,, München, Bavaria
  - Department of Psychiatry and Psychotherapy, Technical University of Munich, University Hospital, München

IPD SHARING:
Plan to Share IPD: Yes
All anonymised study outcomes will be shared, including questionnaire, physiological, and device data.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be made available immediately after the publication of study results, for an unrestricted duration.
Access Criteria: The de-identified individual patient data, i.e., all IPD that underlie results in a publication, will be made accessible after its publication for non-commercial academic projects that have a legitimate research topic and a clearly stated hypothesis. In the event that the application is accepted, researchers will be asked to get the study approved by their institution's ethics board. The study principal investigator will subsequently provide the de-identified data sets via a safe data transfer system.